CLINICAL TRIAL: NCT04799600
Title: The Effect of the Severity of COVID-19 Disease on the Incidence of Acute Renal Failure in ICU
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, ismail aytaç, medical doctor, Ankara City Hospital Bilkent
Other Study IDs: E1-20-1443
Record Dates: First submitted 2021-03-10; First posted 2021-03-16 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: COVID19; Acute Renal Failure
Keywords: COVID19; Acute Renal Failure
MeSH Terms: conditions — COVID-19; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Renal Failure in ICU: COVID-19 Patients with Acute Renal Failure in ICU
  Interventions: Other: BRESCİA-COVİD Respiratory Severity Scale

INTERVENTIONS:
Other: BRESCİA-COVİD Respiratory Severity Scale — KDIGO acute renal failure score BRESCİA-COVID Respiratory Severity Score

SUMMARY:
Aim of the study is to determinate the frequency of acute renal failure in COVID-19 patients, its relationship with the severity of COVID-19 disease in ICU, and the ability to take precautions against these factors.

ELIGIBILITY:
Inclusion Criteria:

Patients hospitalized in the intensive care unit diagnosed with COVID-19 will include in the study.

Exclusion Criteria:

there is no exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in the intensive care unit diagnosed with COVID-19 will participate in the study.
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
KDIGO criteria | 6 months
  KDIGO Criteria stage 1: Increase in SCr by ≥ 0.3 mg/dL within 48 hours or increase in SCr 1.5 to 1.9 times baseline which is known or presumed to have occurred within the prior 7 days Stage 2: 2.0 to 2.9 multiplied by baseline SCr;
  Stage 3: 3.0 or more multiplied by baseline; increase in SCr ≥ 4.0 mg/dL; or beginning of renal replacement therapy regardless of a previous KDIGO stage.
BRESCIA-COVID RESPIRATORY SEVERITY SCALE (BCRSS) scores | 6 months
  The BCRSS score (between level 0-8) is calculated from "www.mdcalc.com/brescia-covid-respiratory-severity-scale-bcrss-algorithm" according to the severity of COVID disease , respiratory rate, PaO2 level, chest x-ray, and clinical status.

CONTACTS AND LOCATIONS:
Overall Officials: betül aytaç, MD, Principal Investigator — ankara ch bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kellum JA, Lameire N; KDIGO AKI Guideline Work Group. Diagnosis, evaluation, and management of acute kidney injury: a KDIGO summary (Part 1). Crit Care. 2013 Feb 4;17(1):204. doi: 10.1186/cc11454. PMID 23394211
- [Result] Wang L, Li X, Chen H, Yan S, Li D, Li Y, Gong Z. Coronavirus Disease 19 Infection Does Not Result in Acute Kidney Injury: An Analysis of 116 Hospitalized Patients from Wuhan, China. Am J Nephrol. 2020;51(5):343-348. doi: 10.1159/000507471. Epub 2020 Mar 31. PMID 32229732
- [Result] Rodriguez-Nava G, Yanez-Bello MA, Trelles-Garcia DP, Chung CW, Friedman HJ, Hines DW. Performance of the quick COVID-19 severity index and the Brescia-COVID respiratory severity scale in hospitalized patients with COVID-19 in a community hospital setting. Int J Infect Dis. 2021 Jan;102:571-576. doi: 10.1016/j.ijid.2020.11.003. Epub 2020 Nov 9. PMID 33181332